

Title: Special Drug Use Surveillance of Leuplin PRO for Injection Kit 22.5 mg for "Prostate Cancer"

NCT Number: NCT03209492

Statistical analysis plan Approve Date: 30-Jan-2018

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

### Statistical Analysis Plan

(Analyses for final tabulation)

Product name : Leuplin PRO for Injection Kit 22.5 mg

Surveillance name : Special drug use surveillance for "prostate cancer"

Protocol number : Leuprorelin-5002

Sponsor : Takeda Pharmaceutical Company Limited



### Table of Contents

| 1 | Def | 1111t1 | ons of Terms, etc. | 3 |
|---|---|---|---|---|
| | 1.1 | List | of Terms and Abbreviations | 3 |
| | 1.2 | Ana | ılysis Sets | 5 |
| | 1.3 | Nu | mber of Digits to be Displayed | 5 |
| | 1.4 | Imp | portant Identified Risks, Important Potential Risks, and Important Missing | |
| | | In | formation | 6 |
| | 1.5 | Oth | er Handling | 7 |
| 2 | Number of Surveillance Medical Institutions, Number of Enrolled Patients, and Patient | | | |
| | Cor | npos | ition | 8 |
| | 2.1 | Dis | position of Patients | 8 |
| 3 | Patient Baseline Characteristics | | | 9 |
| | 3.1 | Pat | ent Baseline Characteristics | 9 |
| 4 | Treatment Given | | | |
| | 4.1 | Tre | atment Status of Prostate Cancer Drug Other Than Leuplin PRO | 11 |
| | 4.2 | Tre | atment Status of Leuplin PRO | 11 |
| | 4.3 | Pre | sence or Absence of and Reason for Discontinuation of Observation | 11 |
| 5 | Mat | tters | on Safety | 12 |
| | 5.1 | Occ | currence of Adverse Events and Adverse Drug Reactions/Infections | 12 |
| | 5. | .1.1 | Occurrence of Adverse Events | 12 |
| | 5. | 1.2 | Occurrence of Adverse Drug Reactions/Infections | 13 |
| | 5. | 1.3 | Occurrence of Adverse Events Corresponding to Important Identified Risks, | |
| | | | Important Potential Risks, or Important Missing Information | 14 |
| | 5. | 1.4 | Occurrence of Adverse Drug Reactions/Infections Corresponding to Important | |
| | | | Identified Risks, Important Potential Risks, or Important Missing Information | 15 |
| | 5.2 | Occ | currence of Adverse Events and Adverse Drug Reactions/Infections by Seriousness, | |
| | | Ti | me of Onset, and Outcome | 16 |
| | 5. | .2.1 | Occurrence of Adverse Events by Seriousness, Time of Onset, and Outcome | 16 |
| | 5. | .2.2 | Occurrence of Adverse Drug Reactions/Infections by Seriousness, Time of Onset, | |
| | | | and Outcome | 17 |
| | 5.3 | Occ | currence of Injection Site Reaction Not Unrelated to Leuplin PRO | 19 |
| | 5. | .3.1 | Occurrence of Injection Site Reaction Not Unrelated to Leuplin PRO | 19 |
| | 5. | .3.2 | Detail of Induration Not Unrelated to Leuplin PRO | 19 |
| | 5. | .3.3 | Incidence of Induration Not Unrelated to Leuplin PRO by Factor | 20 |
| | 5.4 | Occ | currence of Adverse Drug Reactions/Infections by Baseline Characteristics and | |
| | | Tr | eatment Given | 21 |

| | 5.4.1 | Occurrence of Adverse Drug Reactions/Infections by Baseline Characteristics and | |
|---|---|---|---|
| | | Treatment Given | 21 |
| | 5.4.2 | Occurrence of Adverse Drug Reactions/Infections by Age Group | 23 |
| | 5.4.3 | Occurrence of Adverse Drug Reactions/Infections by ECOG Performance Status | 23 |
| | 5.4.4 | Occurrence of Adverse Drug Reactions/Infections by Full-Treatment Status of | |
| | | Leuplin PRO | 23 |
| | 5.4.5 | Occurrence of Adverse Drug Reactions/Infections by Injection Site | 23 |
| | 5.4.6 | Occurrence of Adverse Drug Reactions/Infections by Disease Status | 24 |
| | 5.4.7 | Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of | |
| | | Predisposition to Hypersensitivity | 24 |
| | 5.4.8 | Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of | |
| | | Concurrent Renal Impairment | 24 |
| | 5.4.9 | Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of | |
| | | Concurrent Hepatic Impairment | 24 |
| | 5.4.10 | Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of | |
| | | Concurrent Diabetes Mellitus | 25 |
| | 5.4.11 | Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of | |
| | | Concurrent Hypertension | 25 |
| | 5.4.12 | Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of | |
| | | Concurrent Illness | 25 |
| | 5.4.13 | Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of | |
| | | History of Thromboembolism | 26 |
| | 5.4.14 | Occurrence of Adverse Drug Reactions/Infections by BMI | 26 |
| | 5.4.15 | Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of | |
| | | Treatment with LH-RH Agonist or Antagonist Immediately before the Start of | |
| | | Leuplin PRO Treatment | 26 |
| | 5.4.16 | Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of | |
| | | Treatment with Prostate Cancer Drug Other Than LH-RH Agonists or Antagonists | |
| | | Immediately before the Start of Leuplin PRO Treatment | 26 |
| 4 | 5.5 Occ | surrence of Adverse Drug Reactions/Infections in Additional Pharmacovigilance Plan | |
| | (A | ttachment Style 12) | 28 |
| | 5.6 Sun | nmary of Patients in Post-Marketing Surveillance, etc. (Attachment Style 16) | 29 |
| 1 | Attached | table PTs corresponding to risks | 30 |
| His | story of p | reparation (version control) | 33 |

#### 1 Definitions of Terms, etc.

#### 1.1 List of Terms and Abbreviations

- Leuplin PRO: Leuplin PRO for Injection Kit 22.5 mg is abbreviated as Leuplin PRO.
- Adverse drug reaction (ADR), etc.: ADR, etc. is an abbreviation of ADR/infection. ADRs, etc.
  refer to all adverse events (AEs) other than those assessed by the investigator to be not related to
  Leuplin PRO. In this document, "adverse drug reactions/infections" is used in titles, and "ADRs,
  etc." is used in the text and tables.
- Serious adverse event (SAE): A SAE is an adverse event assessed by the investigator to be serious. Events included in the MedDRA code list in Takeda Medically Significant AE List will be handled as serious even if assessed by the investigator to be not serious.
- Causal relationship: An event assessed as not related to Leuplin PRO will be handled as "not related." Events not unrelated to Leuplin PRO in the text and tables refer to all events other than those assessed as not related to Leuplin PRO.
- Summary statistics: Collective term for number of patients, mean, standard deviation, maximum, minimum, and quartiles
- Patient with no CRF collected: Enrolled patient for whom the CRF has not been collected
- Patient with the CRF collected: Enrolled patient for whom the CRF has been collected
- Finalized patient: Patient for whom the CRF has been collected and finalized at least once by data lock point
- Non-finalized patient: Patient for whom the CRF has been collected, but has not been finalized by data lock point
- Age: If the month and day of starting Leuplin PRO treatment is smaller than the month and day of birth, age will be calculated as year of starting Leuplin PRO treatment year of birth 1. If the month and day of starting Leuplin PRO treatment is equal to or greater than the month and day of birth, age will be calculated as year of starting Leuplin PRO treatment year of birth. If the day of birth is unknown, 1 will be used for calculation.
- Time from diagnosis of prostate cancer to patient registration (months):
  - Actual number (units: month) = ("date of patient registration" "date of diagnosis" + 1)/30.44
- BMI (kg/m²): Calculated as body weight (kg)/height (m)² (displayed to one decimal place by rounding)

- Induration: AE with "induration" selected for "Specific symptom (multiple answers allowed)" in the column of [Adverse event: Injection site reaction] in the CRF
- Prostate cancer drug other than luteinizing hormone-releasing hormone (LH-RH) agonists or antagonists
  - Bicalutamide: Drugs with a NHI drug code starting with 4291009
  - Flutamide: Drugs with a NHI drug code starting with 4291005
  - Other: Other drugs not listed above

#### 1.2 Analysis Sets

The analysis set in this surveillance is safety population. This analysis set is defined as described below.

#### • Safety population

In this document, the safety population is defined as all Leuplin PRO-treated patients evaluable for safety with no major protocol violation. Patients for whom the CRF has been collected will be excluded from the safety population if any of the following criteria is met:

- Not treated with Leuplin PRO
- Treatment before the contract period
- Registration 15 days or more after Leuplin PRO treatment
- It is unknown whether the patient experienced an AE

#### 1.3 Number of Digits to be Displayed

#### • Percentage (%)

Proportion of patients with an AE or an ADR, etc. or number of AE or ADR, etc.:

Displayed to two decimal places by rounding

Other:

Displayed to one decimal place by rounding

#### Summary statistics

Mean, median, first quartile, and third quartile:

Displayed to one lower digit than raw data by rounding

Standard deviation:

Displayed to two lower digits than raw data by rounding

Minimum and maximum:

Displayed to the same number of digits as the relevant data

### 1.4 Important Identified Risks, Important Potential Risks, and Important Missing Information

- Important identified risks
  - Injection site reaction: Injection site reaction is defined as the following AEs:
    - HLT code 10022097 [Infusion site reactions]
    - HLT code 10057196 [Administration site reactions NEC]
    - PT code: Refer to [Attached table PTs corresponding to risks].
  - Decreased bone mass density: Decreased bone mass density is defined as the following AEs:
    - SMQ code 20000178 [Osteoporosis/osteopenia (SMQ) narrow]
    - PT code: Refer to [Attached table PTs corresponding to risks].
  - Diabetes mellitus: Diabetes mellitus is defined as the following AEs:
    - SMQ code 20000041 [Hyperglycemia/new onset diabetes mellitus (SMQ) broad]
  - Interstitial lung disease: Interstitial lung disease is defined as the following AEs:
    - SMQ code 20000042 [Interstitial lung disease (SMQ) narrow]
  - Depression: Depression is defined as the following AEs:
    - SMQ code 20000167 [Depression (excl suicide and self injury) (SMQ) narrow]
    - SMQ code 20000037 [Suicide/self-injury (SMQ) narrow]
  - Thromboembolism: Thromboembolism is defined as the following AEs:
    - SMQ code 20000004 [Cardiac failure (SMQ) narrow]
    - SMQ code 20000166 [Conditions associated with central nervous system haemorrhages and cerebrovascular accidents (SMQ) narrow]
    - SMQ code 20000064 [Haemorrhagic cerebrovascular conditions (SMQ) narrow]
    - SMQ code 20000063 [Ischemic central nervous system vascular conditions (SMQ) narrow]
    - SMQ code 20000165 [Cerebrovascular disorders, not specified as haemorrhagic or ischaemic (SMQ) narrow]
    - SMQ code 20000082 [Embolic and thrombotic events, arterial (SMQ) narrow]
    - SMQ code 20000084 [Embolic and thrombotic events, venous (SMQ) narrow]
    - SMQ code 20000083 [Embolic and thrombotic events, vessel type unspecified and mixed arterial and venous (SMQ) narrow]
    - SMQ code 20000047 [Myocardial infarction (SMQ) broad]
    - SMQ code 20000168 [Other ischaemic heart disease (SMQ) broad]

- Pituitary apoplexy: Pituitary apoplexy is defined as the following AEs:
  - PT code: Refer to [Attached table PTs corresponding to risks].
- Hepatic dysfunction/jaundice: Hepatic dysfunction/jaundice is defined as the following AEs:
  - SMQ code 20000009 [Cholestasis and jaundice of hepatic origin (SMQ) narrow]
  - SMQ code 20000013 [Hepatic failure, fibrosis, and cirrhosis and other liver damage-related conditions (SMQ) narrow]
  - SMQ code 20000010 [Hepatitis, non-infectious (SMQ) narrow]
  - SMQ code 20000008 [Liver related investigations, signs and symptoms (SMQ) narrow]
- Cardiac failure: Cardiac failure is defined as the following AEs:
  - SMQ code 20000004 [Cardiac failure (SMQ) narrow]
- Urinary tract obstruction: Urinary tract obstruction is defined as the following AEs:
  - PT code: Refer to [Attached table PTs corresponding to risks].
- Important potential risks
  - Anaphylaxis: Anaphylaxis is defined as the following AEs:
    - SMQ code 20000021 [Anaphylactic reaction (SMQ) narrow]
    - SMQ code 20000071 [Anaphylactic/anaphylactoid shock conditions (SMQ) narrow]
  - Hypertension: Hypertension is defined as the following AEs:
    - SMQ code 20000147 [Hypertension (SMQ) narrow]
- Important missing information: Not applicable

#### 1.5 Other Handling

• Time of onset of AE (or ADR, etc.): Time of onset of AE (or ADR, etc.) will be calculated as date of onset of AE (or ADR, etc.) - start date of Leuplin PRO treatment + 1. If the day of AE (or ADR, etc.) is unknown, 1 will be used for calculation. If an AE (or ADR, etc.) occurs in the same year and month as Leuplin PRO treatment is started, the start date of Leuplin PRO treatment will be used for calculation.

## 2 Number of Surveillance Medical Institutions, Number of Enrolled Patients, and Patient Composition

#### 2.1 Disposition of Patients

Patients included All enrolled patients (enrolled patients)

in analysis:

Analysis items: Enrolled patients

Number of surveillance medical

institutions

Patients with no CRF collected

Reason for failure to collect [Transfer of the investigator during the

observation period, medical reason

for the investigator, other]

Patients with the CRF collected

Non-finalized patients

Finalized patients

Patients excluded from safety

evaluation\*

Reason for exclusion (multiple

tabulation)

[Not treated with Leuplin PRO,

treatment before the contract period,

registration 15 days or more after

Leuplin PRO treatment, it is

unknown whether the patient

experienced an AE]

Patients included in safety evaluation\*

Analysis methods:

For the aforementioned analysis items, analysis will be performed as described

below, and a patient composition diagram will be prepared.

For enrolled patients, the number of surveillance medical institutions will also be calculated. One medical institution with different departments will be counted as

one medical institution.

\* Patients included in safety evaluation refer to the safety population, and patients excluded from safety evaluation refer to patients excluded from the safety population (finalized patients excluded from the safety population here).

(1) Frequency tabulation

#### 3 Patient Baseline Characteristics

#### 3.1 Patient Baseline Characteristics

Patients included Safety population

in analysis:

Analysis items: Age (years) [<60 years, 60-<65 years, 65-<70

years, 70-<75 years, 75-<80 years,

>=80 years]

[<65 years, >=65 years]

Time from diagnosis of prostate cancer

to patient registration (months)

ECOG Performance Status [0, 1, 2, 3, 4]

Disease status [Patient on postoperative adjuvant

therapy, patient with localized

cancer, patient with locally advanced

cancer, patient with metastatic

cancer]

[No, yes, unknown]

Diagnostic category [Outpatient, inpatient]

Presence or absence of predisposition

to hypersensitivity

Presence or absence of concurrent

illness

Detail of concurrent illness (multiple

tabulation)

[No, yes]

[Diabetes mellitus, hypertension, hepatic disease, renal disease,

allergic disease, malignant tumor,

other]

Presence or absence of history of

thromboembolism

istory of [No, yes, unknown]

Detailed history of thromboembolism

(multiple tabulation)

[Myocardial infarction, cerebral infarction, venous thrombosis, pulmonary embolism, other]

Height (cm)

Body weight (kg)

BMI  $(kg/m^2)$  [<18.5, 18.5-<25.0, 25.0-<30.0,

>=30.0, unknown]

Presence or absence of treatment with

LH-RH agonist or antagonist

immediately before the start of Leuplin

[No, yes]

PRO treatment

Disposition of treatment with LH-RH

agonist or antagonist immediately

before the start of Leuplin PRO

treatment

[Leuprorelin acetate 3.75 mg, leuprorelin acetate 11.25 mg,

[Bicalutamide, flutamide, other]

goserelin 3.6 mg, goserelin 10.8 mg,

degarelix acetate]

[No, yes]

Presence or absence of treatment with

prostate cancer drug other than LH-RH

agonists or antagonists immediately

before the start of Leuplin PRO

treatment

Disposition of treatment with prostate

cancer drug other than LH-RH agonists

or antagonists immediately before the

start of Leuplin PRO treatment

(multiple tabulation)

Analysis methods:

For the aforementioned analysis items, frequency tabulation will be performed

for discrete data, and summary statistics will be calculated for continuous data.

#### 4 Treatment Given

#### 4.1 Treatment Status of Prostate Cancer Drug Other Than Leuplin PRO

Patients included Safety population

in analysis:

Analysis items: Presence or absence of treatment with [No, yes]

prostate cancer drug other than Leuplin

**PRO** 

Disposition of treatment with prostate cancer drug other than Leuplin PRO

(multiple tabulation)

Analysis For the aforementioned analysis items, frequency tabulation will be performed.

methods:

#### 4.2 Treatment Status of Leuplin PRO

Patients included Safety population

in analysis:

Analysis items: Full-treatment status of Leuplin PRO [Yes, no]

Injection site [Extensor surface of the upper arm,

deltoid region of the upper arm,

abdomen, buttocks, other]

Analysis For the aforementioned analysis items, frequency tabulation will be performed.

methods:

#### 4.3 Presence or Absence of and Reason for Discontinuation of Observation

Patients included Safety population

in analysis:

Analysis items: Presence or absence of discontinuation [No, yes]

of observation

Reason for discontinuation of [Patient's failure to visit the hospital

observation such as transfer to another hospital,

death, other]

Analysis For the aforementioned analysis items, frequency tabulation will be performed.

methods:

#### 5 Matters on Safety

#### 5.1 Occurrence of Adverse Events and Adverse Drug Reactions/Infections

#### 5.1.1 Occurrence of Adverse Events

Patients included Safety population

in analysis:

Analysis item: AEs

Analysis For the aforementioned analysis item, analysis will be performed as described

methods: below.

(1) Number of patients with an AE

- (2) Number of AE
- (3) Proportion of patients with an AE
- (4) Type of AE

For each analysis, events or patients will be counted as described below.

[Number of patients with an AE]

• Number of patients who experienced an AE

[Number of AE]

• Number of reported AE. Multiple episodes of the same AE in the same patient will be tabulated as the total number of episodes.

[Proportion of patients with an AE]

• The proportion of patients with an AE will be calculated as number of patients with an AE/number of patients included in safety evaluation × 100.

#### [Type of AE]

- AEs will be coded using the MedDRA/J. AEs will be classified by SOC and then tabulated by PT. For the SOC of investigations, AEs will be sorted by HLGT (lined up in ascending order of HLGT code, but not output) and then tabulated by PT.
- For SOC, the number and proportion of patients with an AE will be listed in internationally agreed SOC order. Multiple episodes of the same SOC in the same patient will be counted as 1 patient for the relevant SOC.
- For PT, the number and proportion of patients with an AE will be listed in ascending order of PT code. Multiple episodes of the same PT in the same patient will be counted as 1 patient for the relevant PT.

#### 5.1.2 Occurrence of Adverse Drug Reactions/Infections

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Analysis For the aforementioned analysis item, analysis will be performed as described

methods: below.

(1) Number of patients with an ADR, etc.

- (2) Number of ADR, etc.
- (3) Incidence of ADR, etc.
- (4) Type of ADR, etc.

For each analysis, events or patients will be counted as described below.

[Number of patients with an ADR, etc.]

• Number of patients who experienced an ADR, etc.

[Number of ADR, etc.]

• Number of reported ADR, etc. Multiple episodes of the same ADR, etc. in the same patient will be tabulated as the total number of episodes.

[Incidence of ADR, etc.]

• The incidence of ADR, etc. will be calculated as number of patients with an ADR, etc./number of patients included in safety evaluation × 100.

[Type of ADR, etc.]

- ADRs, etc. will be coded using the MedDRA/J. ADRs, etc. will be classified by SOC and then tabulated by PT. For the SOC of investigations, ADRs, etc. will be sorted by HLGT (lined up in ascending order of HLGT code, but not output) and then tabulated by PT.
- For SOC, the number and incidence of ADR, etc. will be listed in internationally agreed SOC order. Multiple episodes of the same SOC in the same patient will be counted as 1 patient for the relevant SOC.
- For PT, the number and incidence of ADR, etc. will be listed in ascending order of PT code. Multiple episodes of the same PT in the same patient will be counted as 1 patient for the relevant PT.

## 5.1.3 Occurrence of Adverse Events Corresponding to Important Identified Risks, Important Potential Risks, or Important Missing Information

Patients included Safety population

in analysis:

Analysis item: AEs corresponding to important identified risks, important potential risks, or

important missing information (described in Section 1.4 in Section 1,

"Definitions of Terms, etc.")

Analysis For the aforementioned analysis item, analysis will be performed as described

methods: below.

(1) Number of patients with an AE

- (2) Number of AE
- (3) Proportion of patients with an AE
- (4) Type of AE

For each analysis, events or patients will be counted as described below.

[Number of patients with an AE]

Number of patients who experienced an AE

[Number of AE]

• Number of reported AE. Multiple episodes of the same AE in the same patient will be tabulated as the total number of episodes.

[Proportion of patients with an AE]

• The proportion of patients with an AE will be calculated as number of patients with an AE/number of patients included in safety evaluation × 100.

[Type of AE]

- AEs will be coded using the MedDRA/J. AEs will be classified by SOC and then tabulated by PT. For the SOC of investigations, AEs will be sorted by HLGT (lined up in ascending order of HLGT code, but not output) and then tabulated by PT.
- For SOC, the number and proportion of patients with an AE will be listed in internationally agreed SOC order. Multiple episodes of the same SOC in the same patient will be counted as 1 patient for the relevant SOC.
- For PT, the number and proportion of patients with an AE will be listed in ascending order of PT code. Multiple episodes of the same PT in the same patient will be counted as 1 patient for the relevant PT.

# 5.1.4 Occurrence of Adverse Drug Reactions/Infections Corresponding to Important Identified Risks, Important Potential Risks, or Important Missing Information

Patients included Safety population

in analysis:

Analysis item: ADRs, etc. corresponding to important identified risks, important potential risks,

or important missing information (described in Section 1.4 in Section 1,

"Definitions of Terms, etc.")

Analysis For the aforementioned analysis item, analysis will be performed as described

methods: below.

(1) Number of patients with an ADR, etc.

- (2) Number of ADR, etc.
- (3) Incidence of ADR, etc.
- (4) Type of ADR, etc.

For each analysis, events or patients will be counted as described below.

[Number of patients with an ADR, etc.]

• Number of patients who experienced an ADR, etc.

[Number of ADR, etc.]

• Number of reported ADR, etc. Multiple episodes of the same ADR, etc. in the same patient will be tabulated as the total number of episodes.

[Incidence of ADR, etc.]

• The incidence of ADR, etc. will be calculated as number of patients with an ADR, etc./number of patients included in safety evaluation × 100.

[Type of ADR, etc.]

- ADRs, etc. will be coded using the MedDRA/J. ADRs, etc. will be classified by SOC and then tabulated by PT. For the SOC of investigations, ADRs, etc. will be sorted by HLGT (lined up in ascending order of HLGT code, but not output) and then tabulated by PT.
- For SOC, the number and incidence of ADR, etc. will be listed in internationally agreed SOC order. Multiple episodes of the same SOC in the same patient will be counted as 1 patient for the relevant SOC.
- For PT, the number and incidence of ADR, etc. will be listed in ascending order of PT code. Multiple episodes of the same PT in the same patient will be counted as 1 patient for the relevant PT.

### 5.2 Occurrence of Adverse Events and Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and Outcome

#### 5.2.1 Occurrence of Adverse Events by Seriousness, Time of Onset, and Outcome

Patients included Safety population

in analysis:

Analysis item: AEs
Stratification Total

factors: Seriousness [Serious, not serious]

Time of onset [<7 days, 7-<28 days, 28-<56 days,

56-<84 days, 84-<168 days, >=168

days]

Outcome [Recovered, recovering, not recovered,

recovered with sequelae, died,

unknown, unknown]

Analysis methods:

For the aforementioned analysis item, analysis will be performed in each stratum of the stratification factor as described below.

- (1) Number of patients with an AE
- (2) Number of AE
- (3) Proportion of patients with an AE
- (4) Type of AE

For each analysis, events or patients will be counted as described below.

[Number of patients with an AE]

• Number of patients who experienced an AE

[Number of AE]

• Number of reported AE. Multiple episodes of the same AE in the same patient will be tabulated as the total number of episodes.

[Proportion of patients with an AE]

• The proportion of patients with an AE will be calculated as number of patients with an AE/number of patients included in safety evaluation × 100.

[Type of AE]

- AEs will be coded using the MedDRA/J. AEs will be classified by SOC and then tabulated by PT. For the SOC of investigations, AEs will be sorted by HLGT (lined up in ascending order of HLGT code, but not output) and then tabulated by PT.
- For SOC, the number and proportion of patients with an AE will be listed in internationally agreed SOC order. Multiple episodes of the same SOC in the

same patient will be counted as 1 patient for the relevant SOC. Multiple episodes of the same SOC will be employed as 1 event according to the order of precedence described at the end.

 For PT, the number and proportion of patients with an AE will be listed in ascending order of PT code. Multiple episodes of the same PT in the same patient will be counted as 1 patient for the relevant PT. Multiple episodes of the same PT will be employed as 1 event according to the following order of precedence:

Seriousness: serious → not serious

Time of onset: <7 days  $\rightarrow$  7-<28 days  $\rightarrow$  28-<56 days  $\rightarrow$  56-<84 days  $\rightarrow$ 

84-<168 days  $\rightarrow >=168$  days

Outcome: died  $\rightarrow$  recovered with sequelae  $\rightarrow$  not recovered  $\rightarrow$  recovering

 $\rightarrow$  recovered  $\rightarrow$  unknown

### 5.2.2 Occurrence of Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and Outcome

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Total

factors: Seriousness [Serious, not serious]

Time of onset [<7 days, 7-<28 days, 28-<56 days,

56-<84 days, 84-<168 days, >=168

days]

Outcome [Recovered, recovering, not recovered,

recovered with sequelae, died,

unknown, unknown]

Analysis methods:

For the aforementioned analysis item, analysis will be performed in each stratum of the stratification factor as described below.

- (1) Number of patients with an ADR, etc.
- (2) Number of ADR, etc.
- (3) Incidence of ADR, etc.
- (4) Type of ADR, etc.

For each analysis, events or patients will be counted as described below.

[Number of patients with an ADR, etc.]

• Number of patients who experienced an ADR, etc.

[Number of ADR, etc.]

• Number of reported ADR, etc. Multiple episodes of the same ADR, etc. in the same patient will be tabulated as the total number of episodes.

#### [Incidence of ADR, etc.]

• The incidence of ADR, etc. will be calculated as number of patients with an ADR, etc./number of patients included in safety evaluation × 100.

#### [Type of ADR, etc.]

- ADRs, etc. will be coded using the MedDRA/J. ADRs, etc. will be classified by SOC and then tabulated by PT. For the SOC of investigations, ADRs, etc. will be sorted by HLGT (lined up in ascending order of HLGT code, but not output) and then tabulated by PT.
- For SOC, the number and incidence of ADR, etc. will be listed in
  internationally agreed SOC order. Multiple episodes of the same SOC in the
  same patient will be counted as 1 patient for the relevant SOC. Multiple
  episodes of the same SOC will be employed as 1 event according to the
  order of precedence described at the end.
- For PT, the number and incidence of ADR, etc. will be listed in ascending order of PT code. Multiple episodes of the same PT in the same patient will be counted as 1 patient for the relevant PT. Multiple episodes of the same PT will be employed as 1 event according to the following order of precedence:

Seriousness: serious  $\rightarrow$  not serious

Time of onset: <7 days  $\rightarrow$  7-<28 days  $\rightarrow$  28-<56 days  $\rightarrow$  56-<84 days  $\rightarrow$  84-<168 days  $\rightarrow$  >=168 days

Outcome: died  $\rightarrow$  recovered with sequelae  $\rightarrow$  not recovered  $\rightarrow$  recovering  $\rightarrow$  recovered  $\rightarrow$  unknown

#### 5.3 Occurrence of Injection Site Reaction Not Unrelated to Leuplin PRO

#### 5.3.1 Occurrence of Injection Site Reaction Not Unrelated to Leuplin PRO

Patients included Safety population

in analysis:

Analysis item: Injection site reaction not unrelated to Leuplin PRO Stratification Presence or absence of injection site [No, yes]

factors: reaction

Specific symptom (multiple answers [Pain, pruritus, erythema, swelling,

allowed) induration, abscess, ulcer, other]

Analysis For the aforementioned analysis item, frequency tabulation will be performed in

methods: each stratum of the stratification factor.

#### 5.3.2 Detail of Induration Not Unrelated to Leuplin PRO

Patients included Patients in the safety population who experienced induration not unrelated to

in analysis: Leuplin PRO

Analysis items: Seriousness [Serious, not serious]

Abscess/ulcer [No, yes]

Size of induration (longest diameter) [-10 mm, 11-20 mm, 21-30 mm, 31-40

mm, 41 mm-, unknown]

Number of days from Leuplin PRO [<7 days, 7-<28 days, 28-<56 days,

treatment to the day of onset 56-<84 days, 84-<168 days, >=168

days]

Cause of discontinuation of Leuplin [Yes, no]

PRO treatment

Presence or absence of intervention [No, yes]

Outcome [Recovered, recovering, not recovered,

recovered with sequelae, died,

unknown, unknown]

Number of days from the day of onset [<7 days, 7-<28 days, 28-<56 days,

to "recovered" or "recovering" 56-<84 days, 84-<168 days, >=168

(frequency tabulation with only days]

patients who recovered or were recovering as the denominator)

Analysis For the aforementioned analysis items, frequency tabulation will be performed

methods: for discrete data, and summary statistics will be calculated for continuous data.

#### 5.3.3 Incidence of Induration Not Unrelated to Leuplin PRO by Factor

Patients included Safety population

in analysis:

Analysis item: Induration not unrelated to Leuplin PRO

Stratification Age (years) [<65 years, 65-<75 years, >=75 years]

factors: BMI  $(kg/m^2)$  [<18.5, 18.5-<25.0, 25.0-<30.0,

>=30.0, unknown]

Full-treatment status of Leuplin PRO [Yes, no]

Injection site [Extensor surface of the upper arm,

deltoid region of the upper arm,

abdomen, buttocks, other]

Presence or absence of predisposition

to hypersensitivity

[No, yes, unknown]

Presence or absence of concurrent

allergic disease

Disposition of allergic disease [Bronchial asthma, pollinosis, allergic

[No, yes]

[No, yes]

rhinitis, allergic dermatitis]

Presence or absence of treatment with

LH-RH agonist or antagonist

immediately before the start of Leuplin

PRO treatment

Disposition of treatment with LH-RH [Leuprorelin acetate 3.75 mg, agonist or antagonist immediately leuprorelin acetate 11.25 mg,

before the start of Leuplin PRO goserelin 3.6 mg, goserelin 10.8 mg,

treatment degarelix acetate]

Analysis For the aforementioned analysis item, analysis will be performed in each stratum

methods: of the stratification factor as described below.

(1) Number of patients with induration not unrelated to Leuplin PRO and incidence of induration not unrelated to Leuplin PRO

### 5.4 Occurrence of Adverse Drug Reactions/Infections by Baseline Characteristics and Treatment Given

## 5.4.1 Occurrence of Adverse Drug Reactions/Infections by Baseline Characteristics and Treatment Given

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Age (years) [<65 years, >=65 years]

factors: [<65 years, 65-<75 years, >=75 years]

ECOG Performance Status [0, 1, 2, 3, 4]

Full-treatment status of Leuplin PRO [Yes, no]

Injection site [Extensor surface of the upper arm,

deltoid region of the upper arm,

abdomen, buttocks, other]

[Patient on postoperative adjuvant therapy, patient with localized

cancer, patient with locally advanced

cancer, patient with metastatic

cancer]

Presence or absence of predisposition [No, yes, unknown]

to hypersensitivity

Disease status

Presence or absence of concurrent [No, yes]

renal impairment

Presence or absence of concurrent [No, yes]

hepatic impairment

Presence or absence of concurrent [No, yes]

diabetes mellitus

Presence or absence of concurrent [No, yes]

hypertension

Presence or absence of concurrent [No, yes]

illness

Presence or absence of history of [No, yes, unknown]

thromboembolism

BMI (kg/m<sup>2</sup>) [<18.5, 18.5-<25.0, 25.0-<30.0,

>=30.0, unknown]

Presence or absence of treatment with [No, yes]

LH-RH agonist or antagonist

immediately before the start of Leuplin

PRO treatment

Presence or absence of treatment with [No, yes]

prostate cancer drug other than LH-RH agonists or antagonists immediately

before the start of Leuplin PRO

treatment

Analysis For the aforementioned analysis item, analysis will be performed in each stratum

methods: of the stratification factor as described below.

(1) Number of patients with an ADR, etc. and incidence of ADR, etc.

#### 5.4.2 Occurrence of Adverse Drug Reactions/Infections by Age Group

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Age (years) [<65 years, >=65 years]

factor: [<65 years, 65-<75 years, >=75 years]

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

#### 5.4.3 Occurrence of Adverse Drug Reactions/Infections by ECOG Performance Status

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification ECOG Performance Status [0, 1, 2, 3, 4]

factor:

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

### 5.4.4 Occurrence of Adverse Drug Reactions/Infections by Full-Treatment Status of Leuplin PRO

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Full-treatment status of Leuplin PRO [Yes, no]

factor:

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

#### 5.4.5 Occurrence of Adverse Drug Reactions/Infections by Injection Site

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Injection site [Extensor surface of the upper arm,

factor: deltoid region of the upper arm,

abdomen, buttocks, other]

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

#### 5.4.6 Occurrence of Adverse Drug Reactions/Infections by Disease Status

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Disease status [Patient on postoperative adjuvant

factor: therapy, patient with localized

cancer, patient with locally advanced

cancer, patient with metastatic

cancer]

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

# 5.4.7 Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of Predisposition to Hypersensitivity

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Presence or absence of predisposition [No, yes, unknown]

factor: to hypersensitivity

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

### 5.4.8 Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of Concurrent Renal Impairment

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Presence or absence of concurrent [No, yes]

factor: renal impairment

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

# 5.4.9 Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of Concurrent Hepatic Impairment

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Presence or absence of concurrent [No, yes]

factor: hepatic impairment

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

### **5.4.10** Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of

#### **Concurrent Diabetes Mellitus**

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Presence or absence of concurrent [No, yes]

factor: diabetes mellitus

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

#### 5.4.11 Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of

#### **Concurrent Hypertension**

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Presence or absence of concurrent [No, yes]

factor: hypertension

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

#### 5.4.12 Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of

#### **Concurrent Illness**

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Presence or absence of concurrent [No, yes]

factor: illness

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

### 5.4.13 Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of History of Thromboembolism

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Presence or absence of history of [No, yes, unknown]

factor: thromboembolism

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

#### 5.4.14 Occurrence of Adverse Drug Reactions/Infections by BMI

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.
Stratification BMI (kg/m²)

[<18.5, 18.5-<25.0, 25.0-<30.0,

factor: >=30.0, unknown]

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

# 5.4.15 Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of Treatment with LH-RH Agonist or Antagonist Immediately before the Start of Leuplin PRO Treatment

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Presence or absence of treatment with [No, yes]

factor: LH-RH agonist or antagonist

immediately before the start of Leuplin

PRO treatment

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

# 5.4.16 Occurrence of Adverse Drug Reactions/Infections by Presence or Absence of Treatment with Prostate Cancer Drug Other Than LH-RH Agonists or Antagonists Immediately before the Start of Leuplin PRO Treatment

Patients included Safety population

in analysis:

Analysis item: ADRs, etc.

Stratification Presence or absence of treatment with [No, yes]

factor: prostate cancer drug other than LH-RH

agonists or antagonists immediately before the start of Leuplin PRO

treatment

Analysis For the aforementioned analysis item, analysis as described in Section 5.1.2 will

methods: be performed in each stratum of the stratification factor.

# 5.5 Occurrence of Adverse Drug Reactions/Infections in Additional Pharmacovigilance Plan (Attachment Style 12)

Patients included Safety population

in analysis:

Analysis item: ADRs, etc. corresponding to important identified risks or important potential

risks (described in Section 1.4 in Section 1, "Definitions of Terms, etc.")

Stratification Seriousness [Serious, non-serious]

factor:

Analysis For the aforementioned analysis item, analysis will be performed in each stratum

methods: of the stratification factor as described below in accordance with Notes 1 to 4 in

Attachment style 12 in Notification concerning re-examination, PSEHB/PAB/ED

Notification No. 1128-2 dated 28 November 2017.

(1) Number and proportion of patients with an important identified risk

(2) Number and proportion of patients with an important potential risk

Risk terms and the order of risk terms are specified in Section 1.4 in Section 1,

"Definitions of Terms, etc."

#### 5.6 Summary of Patients in Post-Marketing Surveillance, etc. (Attachment Style 16)

Patients included Patients with the CRF collected

in analysis:

Analysis items: Patient number

Site name

Sex

Date of birth

Reason for use (disease code, disease name)

Concurrent illness (disease code, disease name)

Route of administration

Maximum dose

Mean dose

Units

Duration of use

Concomitant medication (NHI drug code, drug name)

Degree of response

ADR (disease code, disease name, outcome)

CRF number

Dropout

Analysis The aforementioned analysis items will be listed in accordance with Notes 1 to 3

methods: in Attachment style 16 in Notification concerning re-examination,

PSEHB/PAB/ED Notification No. 1128-2 dated 28 November 2017.

### Attached table PTs corresponding to risks

| Risk | PT code | PT |
|----------------|----------|------------------------------------------|
| Injection site | 10022044 | Injection site abscess |
| reaction | 10068791 | Administration site abscess |
| Decreased bone | 10000397 | Acetabulum fracture |
| mass density | 10002544 | Ankle fracture |
| | 10009245 | Clavicle fracture |
| | 10009506 | Closed fracture manipulation |
| | 10010149 | Complicated fracture |
| | 10010214 | Compression fracture |
| | 10014487 | Elevation skull fracture |
| | 10015741 | External fixation of fracture |
| | 10016042 | Facial bones fracture |
| | 10016450 | Femoral neck fracture |
| | 10016454 | Femur fracture |
| | 10016667 | Fibula fracture |
| | 10016970 | Foot fracture |
| | 10016997 | Forearm fracture |
| | 10017076 | Fracture |
| | 10017081 | Fracture delayed union |
| | 10017085 | Fracture malunion |
| | 10017088 | Fracture nonunion |
| | 10017107 | Fracture of clavicle due to birth trauma |
| | 10017290 | Fractured ischium |
| | 10017296 | Fractured maxilla elevation |
| | 10017308 | Fractured sacrum |
| | 10017310 | Fractured skull depressed |
| | 10018720 | Greenstick fracture |
| | 10019114 | Hand fracture |
| | 10020100 | Hip fracture |
| | 10020462 | Humerus fracture |
| | 10021343 | Ilium fracture |
| | 10022576 | Internal fixation of fracture |
| | 10023149 | Jaw fracture |
| | 10028200 | Multiple fractures |
| | 10030527 | Open fracture |

| Risk PT code | | PT |
|--------------|----------|------------------------------------|
| | 10030682 | Open reduction of fracture |
| | 10030684 | Open reduction of spinal fracture |
| | 10031290 | Osteoporotic fracture |
| | 10034122 | Patella fracture |
| | 10034156 | Pathological fracture |
| | 10037802 | Radius fracture |
| | 10039117 | Rib fracture |
| | 10039579 | Scapula fracture |
| | 10040960 | Skull fractured base |
| | 10041541 | Spinal compression fracture |
| | 10041569 | Spinal fracture |
| | 10042015 | Sternal fracture |
| | 10042212 | Stress fracture |
| | 10043827 | Tibia fracture |
| | 10045375 | Ulna fracture |
| | 10048049 | Wrist fracture |
| | 10049164 | Fractured coccyx |
| | 10049514 | Traumatic fracture |
| | 10049946 | Cervical vertebral fracture |
| | 10049947 | Lumbar vertebral fracture |
| | 10049948 | Thoracic vertebral fracture |
| | 10052614 | Comminuted fracture |
| | 10053206 | Fracture displacement |
| | 10053962 | Epiphyseal fracture |
| | 10057147 | Fracture debridement |
| | 10057609 | Fracture reduction |
| | 10059362 | Fractured zygomatic arch elevation |
| | 10061161 | Pelvic fracture |
| | 10061365 | Skull fracture |
| | 10061394 | Upper limb fracture |
| | 10061599 | Lower limb fracture |
| | 10061959 | Fracture treatment |
| | 10066094 | Torus fracture |
| | 10066184 | Avulsion fracture |
| | 10066386 | Impacted fracture |
| | 10069135 | Periprosthetic fracture |

| Risk PT code | | PT |
|---|---|---|
| | 10069723 | Loss of anatomical alignment after fracture reduction |
| | 10070286 | Pubis fracture |
| | 10070884 | Atypical femur fracture |
| | 10072132 | Fracture pain |
| | 10072395 | Atypical fracture |
| | 10073162 | Chance fracture |
| | 10073853 | Osteochondral fracture |
| | 10074362 | Sacroiliac fracture |
| | 10074551 | Limb fracture |
| | 10074807 | Spinal fusion fracture |
| | 10077270 | Surgical fixation of rib fracture |
| | 10077603 | Craniofacial fracture |
| | 10078358 | Costal cartilage fracture |
| | 10078749 | Lisfranc fracture |
| | 10079423 | Fracture blisters |
| | 10079667 | Metaphyseal corner fracture |
| | 10079813 | Fracture infection |
| | 10079864 | Subchondral insufficiency fracture |
| Pituitary apoplexy | 10035092 | Pituitary infarction |
| | 10049760 | Pituitary haemorrhage |
| | 10035104 | Pituitary tumour |
| Urinary tract | 10046555 | Urinary retention |
| obstruction | 10013990 | Dysuria |
| | 10061574 | Urinary tract obstruction |
| | 10059345 | Postrenal failure |
| | 10046459 | Urethral obstruction |
| | 10065584 | Urethral stenosis |
| | 10064895 | Urethral atresia |
| | 10046411 | Ureteric stenosis |
| | 10046399 | Ureteric dilatation |
| | 10046406 | Ureteric dilatation |

### **History of preparation (version control)**

| Version | Date | Person who prepared/changed the SAP | Comment |
|---|---|---|---|
| 1st version | 2018.1.30 | PPD | The 1st version was prepared. |